CLINICAL TRIAL: NCT07226791
Title: A Phase 2 Double-Blind, Placebo-Controlled, Adaptive, Dose-Escalation Study to Evaluate the Safety and Efficacy of AGN-151607-DP (USAN: gemibotulinumtoxinA) for the Achievement of Primary Fascial Closure Without the Use of Component Separation Technique, in Subjects Undergoing Open Abdominal Ventral Hernia Repair
Brief Title: Study of AGN-151607-DP to Assess Adverse Events and Change in Disease Activity in Adult Participants Undergoing Open Abdominal Ventral Hernia Repair
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M24-846
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Ventral Hernia
Keywords: Ventral Hernia; AGN-151607-DP; Primary fascial closure; Open Abdominal Ventral Hernia Repair
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- AGN-151607-DP Dose A (Experimental): Participants will receive AGN-151607-DP Dose A on Day 1.
  Interventions: Drug: AGN-151607-DP
- AGN-151607-DP Dose B (Experimental): Participants will receive AGN-151607-DP Dose B on Day 1.
  Interventions: Drug: AGN-151607-DP
- AGN-151607-DP Dose C (Experimental): Participants will receive AGN-151607-DP Dose C on Day 1.
  Interventions: Drug: AGN-151607-DP
- Placebo for AGN-151607-DP (Placebo Comparator): Participants will receive Placebo for AGN-151607-DP on Day 1.
  Interventions: Drug: Placebo for AGN-151607-DP

INTERVENTIONS:
Drug: AGN-151607-DP — Intramuscular Injection
  Arms: AGN-151607-DP Dose A; AGN-151607-DP Dose B; AGN-151607-DP Dose C
Drug: Placebo for AGN-151607-DP — Intramuscular Injection
  Arms: Placebo for AGN-151607-DP

SUMMARY:
A ventral hernia happens when the muscles in the front of your belly become weak and let abdominal content push through, causing a bulge. If it gets worse, intestines can slip into the bulge, leading to serious pain and health problems. This study aims to asses if AGN-151607-DP is safe and effective for closing the belly wall after open ventral hernia surgery, without needing a complex procedure. Adverse Events and change in disease activity will be assessed.

AGN-151607-DP is an investigational drug being developed to treat ventral hernia. Participants will be randomly placed in treatment groups to receive either AGN151607-DP or matching placebo. Approximately 200 adult participants with midline ventral hernia needing open surgical repair will be enrolled in approximately 30 sites in the United States.

Participants will receive intramuscular injections of AGN-161607-DP or matching placebo on Day 1. Duration of the study is approximately 25 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular weekly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Midline ventral hernia requiring open surgical repair.

Exclusion Criteria:

* Medical condition that may put the participant at increased risk with exposure to AGN-151607-DP, including diagnosed muscular dystrophy (e.g., Duchenne's muscular dystrophy), myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, mitochondrial disease, or any other significant disease which might interfere with neuromuscular function.
* History of abdominal or hernia repair surgery requiring hospitalization within 6 months prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Primary Fascial Closure (PFC) Without Use of Component Separation Technique (CST) in Open Ventral Hernia Surgical Repair | Up to approximately 1 Month
  PFC will be defined as the ability to achieve fascia to fascia midline approximation.
Percentage of Participants Experiencing Adverse Events | Up to approximately 25 Months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving PFC | Up to approximately 1 Month
  PFC will be defined as the ability to achieve fascia to fascia midline approximation.
Percentage of Participants With Usage of CST for the Purpose of PFC | Up to approximately 1 Month
  Percentage of participants with usage of CST will be assessed.
Number of Lateral Abdominal Wall Muscles Released to Achieve PFC | Up to approximately 1 Month
  Number of lateral abdominal wall muscles released to achieve PFC will be assessed.
Change From Baseline in Length of Lateral Abdominal Wall Complex as Measured by Abdominal CT Scan in Supine Position Prior to Surgical Repair | Up to approximately 1 Month
  Change in length of lateral abdominal wall complex will be assessed.
Change From Baseline in Length of Lateral Abdominal Wall Complex as Measured by Abdominal CT Scan Performing Valsalva Maneuver Prior to Surgical Repair | Up to approximately 1 Month
  Change in length of lateral abdominal wall complex will be assessed.
Change From Baseline in Width to the Hernia Defect as Measured by Abdominal CT Scan in Supine Position Prior to Surgical Repair | Up to approximately 1 Month
  Change in width to the hernia defect will be assessed.
Change From Baseline in Width to the Hernia Defect as Measured by Abdominal CT Scan Performing Valsalva Maneuver Prior to Surgical Repair | Up to approximately 1 Month
  Change in width to the hernia defect will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-846